CLINICAL TRIAL: NCT00744068
Title: Four Models of Telephone Support for Stimulant Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01DA018208-01A1 (NIH); R01DA018208 (NIH)
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Drug Addiction
Keywords: Stimulant; Drug treatment; Continuing care; Telephone support; Aftercare
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Structured Directive Telephone Support Calls
  Interventions: Behavioral: Continuing Care Telephone Support
- 2 (Experimental): Structured Non-Directive Telephone Continuing Care Support
  Interventions: Behavioral: Continuing Care Telephone Support
- 3 (Experimental): Unstructured Directive Telephone Support
  Interventions: Behavioral: Continuing Care Telephone Support
- 4 (Experimental): Unstructured Non-Directive Telephone Support
  Interventions: Behavioral: Continuing Care Telephone Support
- 5 (No Intervention)

INTERVENTIONS:
Behavioral: Continuing Care Telephone Support — Counselor-provided telephone support as strategies to promote patient aftercare attendance and sustained abstinence from stimulant use. To this end, we will develop and compare the efficacy of four low-cost telephone support protocols for patients who have completed the intensive phase of a structured, outpatient stimulant abuse treatment program.
  Arms: 1; 2; 3; 4

SUMMARY:
The overall objective of this research is to develop and refine empirically supported continuing care interventions that promote healthy behavior and sustained abstinence from illicit drug use.

DETAILED DESCRIPTION:
For treatment interventions to provide the desired result of long term abstinence, it is important to develop strategies to enhance the effectiveness of continued care approaches. We plan to conduct a prospective, randomized comparison of four models of counselor-provided telephone support as strategies to promote patient aftercare attendance and sustained abstinence from stimulant use. To this end, we will develop and compare the efficacy of four low-cost telephone support protocols for patients who have completed the intensive phase of a structured, outpatient stimulant abuse treatment program. Some 500 participants completing a 4-month Matrix Outpatient Model of stimulant abuse treatment will be randomly assigned to one of four counseling groups (n=100 per group): (1) unstructured/non-directive, (2) structured/non-directive, (3) unstructured/directive, or (4) structured/directive telephone counseling, or (5) a control group consisting of standard referral to Matrix aftercare, for a total sample size of 500. The two structured conditions will be based on the behavioral "prompts" identified by Farabee et al. (2002)* as being associated with drug avoidance. In the non-directive conditions, subjects will be allowed to state their own goals and how they intend to achieve them. In the directive conditions, the counselor will provide specific recommendations to help the subject adopt as many of the drug-avoidance activities as possible. Outcomes will be tracked for 12 months following completion of primary treatment (a total of 16 months after treatment admission) and will include measurement of participation in drug-avoidance activities (including aftercare participation) as well as self-reported and objective measures of substance use and related behavior change.

*Farabee, D., Rawson, R.A., & McCann, M. (2002). Adoption of drug avoidance activities among patients in contingency management and cognitive-behavioral treatments. Journal of Substance Abuse Treatment, 23, 343-350.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, 18-65 years of age.
* Meet DSM-IV criteria (at the time of treatment admission) for cocaine or methamphetamine abuse/dependence.
* Have completed the primary phase of treatment at a Matrix outpatient clinic.
* Have telephone access throughout the study procedures.
* Be able to understand and complete rating scales and to follow instructions.
* Be willing to sign an informed consent form.

Exclusion Criteria:

* Have participated in a treatment-related study conducted by the PI and colleagues during the previous 3 years and/or is currently enrolled in a treatment-related study.
* Have any medical, legal, housing or transportation problem which would preclude either safe or consistent participation.
* Have dropped out of the primary phase of treatment prior to completion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2006-04; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Urinalyses | At 3 months and 12 months
Breathalyzer tests | At 3 months and 12 months
Self-report of drug or alcohol use | At 3 months and 12 months
Amount of Treatment Activities | At 3 months and 12 months
Length of Treatment Episode | At 3 months and 12 months

SECONDARY OUTCOMES:
Addiction Severity Index (ASI) | At 3 months and 12 months
HIV Risk-taking Behavior Scale | At 3 months and 12 months
Concurrent Psychosocial Treatments | At 3 months and 12 months
Drug Avoidance Activities (DAA) Survey | At 3 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Farabee, Ph.D., Principal Investigator — UCLA Integrated Substance Abuse Programs
Locations (6):
- United States (6):
  - Twin Town Treatment Center, Los Alamitos, California
  - Matrix Institute on Addictions, Los Angeles, California
  - UCLA Integrated Substance Abuse Programs, Los Angeles, California
  - Matrix Institute on Addictions, Rancho Cucamonga, California
  - Twin Town Treatment Center, West Hollywood, California
  - Matrix Institute on Addicitions, Woodland Hills, California

REFERENCES:
- [Background] Ahles TA, Schlundt DG, Prue DM, Rychtarik RG. Impact of aftercare arrangements on the maintenance of treatment success in abusive drinkers. Addict Behav. 1983;8(1):53-8. doi: 10.1016/0306-4603(83)90056-4. PMID 6308970
- [Background] Allen K. Barriers to treatment for addicted African-American women. J Natl Med Assoc. 1995 Oct;87(10):751-6. PMID 7473850
- [Background] Ashery RS, Carlson RG, Falck RS, Siegal HA. Injection drug users, crack-cocaine users, and human services utilization: an exploratory study. Soc Work. 1995 Jan;40(1):75-82. PMID 7863375
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Battjes RJ, Onken LS, Delany PJ. Drug abuse treatment entry and engagement: report of a meeting on treatment readiness. J Clin Psychol. 1999 May;55(5):643-57. doi: 10.1002/(sici)1097-4679(199905)55:53.0.co;2-s. PMID 10392794
- [Background] Brown BS, O'Grady KE, Battjes RJ, Farrell EE, Smith NP, Nurco DN. Effectiveness of a stand-alone aftercare program for drug-involved offenders. J Subst Abuse Treat. 2001 Dec;21(4):185-92. doi: 10.1016/s0740-5472(01)00201-x. PMID 11777667
- [Background] Burton P, Gurrin L, Sly P. Extending the simple linear regression model to account for correlated responses: an introduction to generalized estimating equations and multi-level mixed modelling. Stat Med. 1998 Jun 15;17(11):1261-91. doi: 10.1002/(sici)1097-0258(19980615)17:113.0.co;2-z. PMID 9670414
- [Background] De Leon G, Melnick G, Kressel D, Jainchill N. Circumstances, motivation, readiness, and suitability (the CMRS scales): predicting retention in therapeutic community treatment. Am J Drug Alcohol Abuse. 1994 Nov;20(4):495-515. doi: 10.3109/00952999409109186. PMID 7832182
- [Background] De Leon G, Melnick G, Thomas G, Kressel D, Wexler HK. Motivation for treatment in a prison-based therapeutic community. Am J Drug Alcohol Abuse. 2000 Feb;26(1):33-46. doi: 10.1081/ada-100100589. PMID 10718162
- [Background] Dees SM, Dansereau DF, Peel JL, Boatler JG, Knight K. Using conceptual matrices, knowledge maps, and scripted cooperation to improve personal management strategies. J Drug Educ. 1991;21(3):211-30. doi: 10.2190/KJKM-F0UR-RDPH-8NUK. PMID 1919960
- [Background] Diez-Roux AV. Multilevel analysis in public health research. Annu Rev Public Health. 2000;21:171-92. doi: 10.1146/annurev.publhealth.21.1.171. PMID 10884951
- [Background] Farabee D, Rawson R, McCann M. Adoption of drug avoidance activities among patients in contingency management and cognitive-behavioral treatments. J Subst Abuse Treat. 2002 Dec;23(4):343-50. doi: 10.1016/s0740-5472(02)00297-0. PMID 12495796
- [Background] Fischer B, Chin AT, Kuo I, Kirst M, Vlahov D. Canadian illicit opiate users' views on methadone and other opiate prescription treatment: an exploratory qualitative study. Subst Use Misuse. 2002 Mar;37(4):495-522. doi: 10.1081/ja-120002807. PMID 12064431
- [Background] Fitzgerald JL, Mulford HA. An experimental test of telephone aftercare contacts with alcoholics. J Stud Alcohol. 1985 Sep;46(5):418-24. doi: 10.15288/jsa.1985.46.418. PMID 2999514
- [Background] Fortney JC, Booth BM, Blow FC, Bunn JY. The effects of travel barriers and age on the utilization of alcoholism treatment aftercare. Am J Drug Alcohol Abuse. 1995 Aug;21(3):391-406. doi: 10.3109/00952999509002705. PMID 7484987
- [Background] Haynes RB, McDonald HP, Garg AX. Helping patients follow prescribed treatment: clinical applications. JAMA. 2002 Dec 11;288(22):2880-3. doi: 10.1001/jama.288.22.2880. PMID 12472330
- [Background] Huber A, Lord RH, Gulati V, Marinelli-Casey P, Rawson R, Ling W. The CSAT methamphetamine treatment program: research design accommodations for "real world" application. J Psychoactive Drugs. 2000 Apr-Jun;32(2):149-56. doi: 10.1080/02791072.2000.10400223. PMID 10908002
- [Background] Huber A, Ling W, Shoptaw S, Gulati V, Brethen P, Rawson R. Integrating treatments for methamphetamine abuse: a psychosocial perspective. J Addict Dis. 1997;16(4):41-50. doi: 10.1080/10550889709511142. PMID 9328808
- [Background] Hunt WA, Barnett LW, Branch LG. Relapse rates in addiction programs. J Clin Psychol. 1971 Oct;27(4):455-6. doi: 10.1002/1097-4679(197110)27:43.0.co;2-r. No abstract available. PMID 5115648
- [Background] Hser YI, Anglin D, Powers K. A 24-year follow-up of California narcotics addicts. Arch Gen Psychiatry. 1993 Jul;50(7):577-84. doi: 10.1001/archpsyc.1993.01820190079008. PMID 8317951
- [Background] Hser YI, Hoffman V, Grella CE, Anglin MD. A 33-year follow-up of narcotics addicts. Arch Gen Psychiatry. 2001 May;58(5):503-8. doi: 10.1001/archpsyc.58.5.503. PMID 11343531
- [Background] Iguchi MY, Belding MA, Morral AR, Lamb RJ, Husband SD. Reinforcing operants other than abstinence in drug abuse treatment: an effective alternative for reducing drug use. J Consult Clin Psychol. 1997 Jun;65(3):421-8. doi: 10.1037//0022-006x.65.3.421. PMID 9170765
- [Background] Intagliata J. A telephone follow-up procedure for increasing the effectiveness of a treatment program for alcoholics. J Stud Alcohol. 1976 Sep;37(9):1330-5. doi: 10.15288/jsa.1976.37.1330. PMID 185468
- [Background] Karno MP, Beutler LE, Harwood TM. Interactions between psychotherapy procedures and patient attributes that predict alcohol treatment effectiveness: a preliminary report. Addict Behav. 2002 Sep-Oct;27(5):779-97. doi: 10.1016/s0306-4603(01)00209-x. PMID 12201384
- [Background] Koumans AJ, Muller JJ, Miller CF. Use of telephone calls to increase motivation for treatment in alcoholics. Psychol Rep. 1967 Aug;21(1):327-8. doi: 10.2466/pr0.1967.21.1.327. No abstract available. PMID 6078383
- [Background] Lash SJ, Blosser SL. Increasing adherence to substance abuse aftercare group therapy. J Subst Abuse Treat. 1999 Jan;16(1):55-60. doi: 10.1016/s0740-5472(98)00015-4. PMID 9888122
- [Background] Lash SJ, Dillard W. Encouraging participation in aftercare group therapy among substance-dependent men. Psychol Rep. 1996 Oct;79(2):585-6. doi: 10.2466/pr0.1996.79.2.585. PMID 8909084
- [Background] Lovejoy M, Rosenblum A, Magura S, Foote J, Handelsman L, Stimmel B. Patients' perspective on the process of change in substance abuse treatment. J Subst Abuse Treat. 1995 Jul-Aug;12(4):269-82. doi: 10.1016/0740-5472(95)00027-3. PMID 8830154
- [Background] MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychol Methods. 2002 Mar;7(1):83-104. doi: 10.1037/1082-989x.7.1.83. PMID 11928892
- [Background] McDonald HP, Garg AX, Haynes RB. Interventions to enhance patient adherence to medication prescriptions: scientific review. JAMA. 2002 Dec 11;288(22):2868-79. doi: 10.1001/jama.288.22.2868. PMID 12472329
- [Background] McKay JR. Effectiveness of continuing care interventions for substance abusers. Implications for the study of long-term treatment effects. Eval Rev. 2001 Apr;25(2):211-32. doi: 10.1177/0193841X0102500205. PMID 11317717
- [Background] McKay JR, McLellan AT, Alterman AI, Cacciola JS, Rutherford MJ, O'Brien CP. Predictors of participation in aftercare sessions and self-help groups following completion of intensive outpatient treatment for substance abuse. J Stud Alcohol. 1998 Mar;59(2):152-62. doi: 10.15288/jsa.1998.59.152. PMID 9500302
- [Background] Pan W. Sample size and power calculations with correlated binary data. Control Clin Trials. 2001 Jun;22(3):211-27. doi: 10.1016/s0197-2456(01)00131-3. PMID 11384786
- [Background] Peterson KA, Swindle RW, Phibbs CS, Recine B, Moos RH. Determinants of readmission following inpatient substance abuse treatment: a national study of VA programs. Med Care. 1994 Jun;32(6):535-50. doi: 10.1097/00005650-199406000-00001. PMID 8189773
- [Background] Ouimette PC, Moos RH, Finney JW. Influence of outpatient treatment and 12-step group involvement on one-year substance abuse treatment outcomes. J Stud Alcohol. 1998 Sep;59(5):513-22. doi: 10.15288/jsa.1998.59.513. PMID 9718103
- [Background] Rawson RA, Shoptaw SJ, Obert JL, McCann MJ, Hasson AL, Marinelli-Casey PJ, Brethen PR, Ling W. An intensive outpatient approach for cocaine abuse treatment. The Matrix model. J Subst Abuse Treat. 1995 Mar-Apr;12(2):117-27. doi: 10.1016/0740-5472(94)00080-b. PMID 7623389
- [Background] Rawson RA, Marinelli-Casey P, Anglin MD, Dickow A, Frazier Y, Gallagher C, Galloway GP, Herrell J, Huber A, McCann MJ, Obert J, Pennell S, Reiber C, Vandersloot D, Zweben J; Methamphetamine Treatment Project Corporate Authors. A multi-site comparison of psychosocial approaches for the treatment of methamphetamine dependence. Addiction. 2004 Jun;99(6):708-17. doi: 10.1111/j.1360-0443.2004.00707.x. PMID 15139869
- [Background] Rawson RA, Obert JL, McCann MJ, Ling W. Neurobehavioral treatment for cocaine dependency: a preliminary evaluation. NIDA Res Monogr. 1993;135:92-115. PMID 8289906
- [Background] Richter KP, Bammer G. A hierarchy of strategies heroin-using mothers employ to reduce harm to their children. J Subst Abuse Treat. 2000 Dec;19(4):403-13. doi: 10.1016/s0740-5472(00)00137-9. PMID 11166505
- [Background] Rochon J. Application of GEE procedures for sample size calculations in repeated measures experiments. Stat Med. 1998 Jul 30;17(14):1643-58. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-3. PMID 9699236
- [Background] Shoptaw S, Rawson RA, McCann MJ, Obert JL. The Matrix model of outpatient stimulant abuse treatment: evidence of efficacy. J Addict Dis. 1994;13(4):129-41. doi: 10.1300/j069v13n04_02. PMID 7734464
- [Background] Shrout PE, Bolger N. Mediation in experimental and nonexperimental studies: new procedures and recommendations. Psychol Methods. 2002 Dec;7(4):422-45. PMID 12530702
- [Background] Silverman K, Higgins ST, Brooner RK, Montoya ID, Cone EJ, Schuster CR, Preston KL. Sustained cocaine abstinence in methadone maintenance patients through voucher-based reinforcement therapy. Arch Gen Psychiatry. 1996 May;53(5):409-15. doi: 10.1001/archpsyc.1996.01830050045007. PMID 8624184
- [Background] Sobell LC, Maisto SA, Sobell MB, Cooper AM. Reliability of alcohol abusers' self-reports of drinking behavior. Behav Res Ther. 1979;17(2):157-60. doi: 10.1016/0005-7967(79)90025-1. No abstract available. PMID 426744
- [Background] Spitzer RL, Williams JB, Gibbon M, First MB. The Structured Clinical Interview for DSM-III-R (SCID). I: History, rationale, and description. Arch Gen Psychiatry. 1992 Aug;49(8):624-9. doi: 10.1001/archpsyc.1992.01820080032005. PMID 1637252
- [Background] Stahler GJ, Cohen E. Using ethnographic methodology in substance abuse treatment outcome research. J Subst Abuse Treat. 2000 Jan;18(1):1-8. doi: 10.1016/s0740-5472(99)00029-x. PMID 10636600
- [Background] Stout RL, Wirtz PW, Carbonari JP, Del Boca FK. Ensuring balanced distribution of prognostic factors in treatment outcome research. J Stud Alcohol Suppl. 1994 Dec;12:70-5. doi: 10.15288/jsas.1994.s12.70. PMID 7723001
- [Result] Farabee D, Cousins SJ, Brecht ML, Antonini VP, Lee AB, Brummer J, Hemberg J, Karno M, Rawson RA. A comparison of four telephone-based counseling styles for recovering stimulant users. Psychol Addict Behav. 2013 Mar;27(1):223-9. doi: 10.1037/a0029572. Epub 2012 Aug 6. PMID 22867295
- See also: Related Info — http://www.uclaisap.org